CLINICAL TRIAL: NCT03762499
Title: Hypertension Management in Young Adults Personalised by Echocardiography and Clinical Outcome.
Acronym: HyperEcho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 247606
Record Dates: First submitted 2018-11-06; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
Keywords: Young adults; Echocardiography
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective participants (Active Comparator): 250 participants will be recruited prospectively during the hypertension clinic, where a full set of data will be collected from each participant as part of their standard hypertension clinical service. An additional echocardiography scan will be performed for this cohort by the study team, if the scan has not been performed as a part of the clinical care service
  Interventions: Diagnostic Test: Echocardiography scan
- Retrospective participants (No Intervention): 500 participants will be recruited retrospectively, and no additional echocardiography scan will be required for them.

INTERVENTIONS:
Diagnostic Test: Echocardiography scan — Non-invasive ultrasound imaging of the heart.
  Arms: Prospective participants

SUMMARY:
HyperEcho is a multi-centre longitudinal observational study, to investigate whether baseline transthoracic echocardiography along with routine data collected in the hypertension clinic can guide clinicians to better manage, and improve risk stratification for cardiovascular disease in young adults with hypertension. Participants are characterised as young adult patients aged between 18 to 40 years old and referred to the hypertension clinic to manage their blood pressure. The study visit will be carried out during the planned routine visit of the participants to the hypertension clinics of NHS trusts within England. Routine data will be collected by the assigned nurse for the hypertension clinic as part of the clinical service, and research participation will not affect the clinical progress of the participant. The additional research component to the clinic will be asking the participants for their consent to undergo a research echocardiography scan if it has not been a part of their clinical assessment. Participants will also be asked to consent to the use of their data that has been collected in the hypertension clinic, such as; referral letters, medical history, 24-hour blood pressure monitoring report, ECG, blood samples, body fat composition, and dietary questionnaire. In addition to this, participants will be asked to consent to further review of their data and medical notes during their follow up visits (up to 10 years).

DETAILED DESCRIPTION:
HyperEcho is a multi-centre longitudinal observational study, to investigate whether baseline transthoracic echocardiography along with routine data collected in the hypertension clinic can guide clinicians to better manage, and improve risk stratification for cardiovascular disease in young adults with hypertension. Participants are characterised as hypertensive patients aged between 18 to 40 years old and referred to the hypertension clinic to manage their blood pressure. A patient and public involvement exercise has been performed to ensure this study design would appeal to patients attending the hypertension clinic, and to investigate the preferred method of contact.

The study visit will be carried out during the planned routine visit of the participants to the hypertension clinics of NHS trusts within England. Routine data will be collected by the assigned nurse for the hypertension clinic as part of the clinical service, and research participation will not affect the clinical progress of the participant. The additional research component to the clinic will be asking the participants for their consent to undergo a research echocardiography scan if it has not been a part of their clinical assessment. Participants will also be asked to consent to the use of their data that has been collected in the hypertension clinic, such as; referral letters, medical history, 24-hour blood pressure monitoring report, ECG, blood samples, body fat composition, and dietary questionnaire. In addition to this, participants will be asked to consent to further review of their data and medical notes during their follow up visits (up to 10 years).

Previous young adult patients who visited the Hypertension clinics in the last 10 years will be also recruited. This cohort will be asked to consent to allow the research team to collect and use their clinical data as well as follow up their medical notes. They will not actively participate in the study as they will not require visiting the hypertension clinic or undergoing an echocardiography scan.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 - 40 years (at the time of their appointment at the hypertension clinic).
* Referred for a Hypertension Clinic in England.

Exclusion Criteria:

* Unable or unwilling to give valid consent for participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2028-10-02 (Estimated)

PRIMARY OUTCOMES:
Identification of patient clusters based on echocardiographic and clinical findings | Obtained at the first clinical visit
  Number of hypertension patient clusters based on echocardiographic and clinical findings

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Clinical Research Facility, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes